CLINICAL TRIAL: NCT02689492
Title: SATisfaction and Adherence to COPD Treatment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.51
Record Dates: First submitted 2015-11-17; First posted 2016-02-24 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The present study will explore the patients satisfaction to COPD medical treatment (i.e. pharmacological and not pharmacological treatment) in a clinical real-world setting and how the satisfaction for medical treatment is related to clinical parameters, quality of life, illness perception and treatment adherence evolution.

Moreover health care resource consumption will be observed during the observation period.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged equal or more than 40 years
2. Patients must have a documented diagnosis of chronic obstructive pulmonary disease (COPD)
3. Patients with no exacerbations in the last 3 months
4. Patients requiring regular treatment according to GOLD guidelines, i.e.: undergoing stable pharmacological treatment for COPD since at least 3 months
5. Written informed consent to both participation in the study and privacy form
6. Patients capable of discernment and able to read or write in Italian language.

Exclusion criteria:

1. Patients who are currently participating in a clinical trial on experimental drugs.
2. Patients naïve to pharmacological treatment for COPD
3. Diagnosis of Asthma COPD Overlap Syndrome (ACOS)

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD pts
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (20):
- Italy (20):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - I.N.R.C.A. - I.R.C.C.S Ospedale Geriatrico Ugo Sestili, Ancona
  - Ospedale Reg Umberto Parini, Aosta
  - A. O. Giuseppe Moscati, Avellino
  - Ospedale Civile di Battipaglia, Battipaglia Salerno
  - IRCCS - Istituto Scientifico di Cassano delle Murge, Cassano Murge Bari
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, CONA (FE)
  - Policlinico San Martino, Genova
  - Az. Unità Loc. Socio-Sanitaria 21 -, Legnago
  - Spedali Riuniti di Livorno, Livorno
  - Fondazione Salvatore Maugeri, Milan
  - Asst Santi Paolo E Carlo, Milan
  - Osp. dei Colli Monaldi-Cotugno, Napoli
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Unità Sanitaria Locale di Reggio Emilia, Reggio Emilia
  - Pol. Universitario Tor Vergata, Roma
  - Ospedale Civile Mazzini, Teramo
  - ASL 4 di Terni, Terni

REFERENCES:
- [Derived] Contoli M, Rogliani P, Di Marco F, Braido F, Corsico AG, Amici CA, Piro R, Sarzani R, Lessi P, Scognamillo C, Scichilone N, Santus P; SAT Study Group. Satisfaction with chronic obstructive pulmonary disease treatment: results from a multicenter, observational study. Ther Adv Respir Dis. 2019 Jan-Dec;13:1753466619888128. doi: 10.1177/1753466619888128. PMID 31760881
- [Derived] Corsico AG, Braido F, Contoli M, Di Marco F, Rogliani P, Scognamillo C, Olivi I, Santus P, Scichilone N, Lazzaro C. Healthcare costs of the SATisfaction and adherence to COPD treatment (SAT) study follow-up. Respir Med. 2019 Jul;153:68-75. doi: 10.1016/j.rmed.2019.05.017. Epub 2019 May 29. PMID 31174106
- [Derived] Baiardini I, Rogliani P, Santus P, Corsico AG, Contoli M, Scichilone N, Di Marco F, Lessi P, Scognamillo C, Molinengo G, Ferri F, Patella V, Fiorentino G, Carone M, Braido F. Disease awareness in patients with COPD: measurement and extent. Int J Chron Obstruct Pulmon Dis. 2018 Dec 17;14:1-11. doi: 10.2147/COPD.S179784. eCollection 2019. PMID 30587957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, non-interventional (observational), prospective cohort study based mainly on newly-collected data for Chronic obstructive pulmonary disease (COPD) patients. No treatments were administered to the patients on the protocol basis, since this was a non-interventional study. The total number of enrolled patients was 401.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial if any one of the specific entry criteria were not met.
Groups:
- Total COPD Patients: Patients were enrolled (enrollment phase was 10 months) in the SAT (SATisfaction and adherence to COPD treatment) study and they were evaluable for the analyses and follow-up visits were scheduled at 6 and 12 months. All patients had a baseline Treatment Satisfaction Questionnaire- 9 items (TSQM-9) usable for the baseline data analysis and were included in the Full Analysis Set (FAS).
Period: Overall Study
Arm/Group | Total COPD Patients
Started | 401
Completed | 315
Not Completed | 86
Not completed — Lost to Follow-up | 61
Not completed — Withdrawal by Subject | 11
Not completed — Death | 9
Not completed — Physician Decision | 2
Not completed — Withdrawal/Loss To Follow-Up | 1
Not completed — Withdrawal/ Physician's Decision | 1
Not completed — Other than listed | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS includes all enrolled patients evaluable for baseline data analysis.
Arm/Group | Total COPD Patients
Number analyzed (Participants) | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented.
  Years | 71.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female.
  Participants
    Female | 102
    Male | 299
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data. Ethnicity was not captured in this trial.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 400
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Patients' Satisfaction With Chronic Obstructive Pulmonary Disease (COPD) Medical Treatments During a 12-month Observation Period
Description: Patient's self-reported satisfaction or dissatisfaction with pharmacological treatments was measured using the Treatment Satisfaction Questionnaire for Medication (TSQM) Version 1.4, a validated instrument. The TSQM has total 9 items (TSMQ-9) with responses to nearly all items rated on a 5-point or 7-point rating scale that provide scores on 3 scales: effectiveness (items #1 #2 #3), convenience (items #4 #5 #6) and global satisfaction (items #7 #8 #9).
  The TSQM-9 domain scores were calculated as recommended by the instrument authors. (i) Effectiveness = [(item1 + item2 + item3) - 3]/18*100, (ii) Convenience = [(item4 + item5 + item6) - 3]/18*100 and (iii) Global satisfaction = [(item7 + item8 + item9) - 3]/14*100.
  Each domain score can be calculated only if all the three items considered in the calculation of that score are not missing. The TSQM-9 domain scores range from 0 to 100, with higher scores representing higher satisfaction on that domain.
Time Frame: At enrollment visit, 6-month follow-up visit and 12-month follow-up visit.
Population: Full Analysis Set (FAS): FAS includes all enrolled patients evaluable for baseline data analysis.
Measure: Mean (Standard Deviation); unit: Unit on Scale
Groups:
- Enrollment Visit: Long-term data on the patients' satisfaction to COPD medical treatments (i.e. pharmacological and not pharmacological treatment) at the enrollment visit. (FAS patients)
- 6-month Follow-up: Long-term data on the patients' satisfaction to COPD medical treatments (i.e. pharmacological and not pharmacological treatment)evaluable at 6 months.
- 12-month Follow-up: Long-term data on the patients' satisfaction to COPD medical treatments (i.e. pharmacological and not pharmacological treatment)evaluable at 12 months.
Arm/Group | Enrollment Visit | 6-month Follow-up | 12-month Follow-up
Number analyzed (Participants) | 401 | 360 | 308
Unit on Scale
  Effectiveness (0-100): number analyzed (Participants) | 400 | 359 | 304
  Effectiveness (0-100) | 64.2 (17.2) | 66.2 (16.3) | 67.1 (15.1)
  Convenience (0-100): number analyzed (Participants) | 390 | 356 | 304
  Convenience (0-100) | 75.8 (15.9) | 75.7 (15.8) | 76.1 (14.0)
  Global satisfaction (0-100): number analyzed (Participants) | 391 | 355 | 305
  Global satisfaction (0-100) | 65.7 (17.1) | 67.5 (16.9) | 67.3 (15.4)

2. Secondary Outcome: Measurements of Patient Disease Perception, Adherence to COPD Treatment, Health Status and Dyspnea Over 12-months Observation Period.
Description: Patient's disease perception was evaluated by Brief Illness Perception Questionnaire (B-IPQ) consist 8 questionnaires rated 1 - 10 response scale. Mean total score ranges from 8-80, where a greater score indicated a more threatening view of COPD.
  Adherence was measured using Morisky Medication Adherence Scale, 4 items (MMAS-4) questionnaire which consists of 4 questions. Items are summed to give an adherence score ranging from 0 to 4, where a higher score indicated a greater adherence grade.
  Patients' health status was measured using the COPD Assessment Test (CAT) questionnaire that consists of 8-items in which patients can choose a score from 0 to 5. The total score ranges from 0 to 40, where a higher score indicated a worst impact of symptoms on the patient's daily activities.
  Dyspnea was measured using Modified Medical Research Council Dyspnea Scale (MMRC) with a 0-to-4 grading system. It had 0-to-4 grading system, with higher score indicating a higher level of dyspnea.
Time Frame: At enrollment visit, 6-month follow-up visit and 12-month follow-up visit
Population: FAS
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | Enrollment Visit | 6-month Follow-up | 12-month Follow-up
Number analyzed (Participants) | 401 | 360 | 308
Unit on Scale
  B-IPQ (8-80): number analyzed (Participants) | 396 | 351 | 304
  B-IPQ (8-80) | 41.8 (11.3) | 42.0 (10.0) | 42.6 (10.5)
  MMAS-4 (0-4) | 3.4 (0.9) | 3.5 (0.9) | 3.5 (0.9)
  CAT score (0-40): number analyzed (Participants) | 401 | 360 | 307
  CAT score (0-40) | 15.7 (7.8) | 15.9 (7.6) | 15.1 (7.5)
  Patients' dyspnea (MMRC): number analyzed (Participants) | 400 | 358 | 305
  Patients' dyspnea (MMRC) | 1.6 (1.1) | 1.8 (1.1) | 1.7 (1.1)

3. Secondary Outcome: The Relationship Between Treatment Satisfaction - Effectiveness Domain and Demographics, Clinical Parameters and Patient Reported Outcome (PROs) During a 12-month Observation Period.
Description: A regression model was estimated, where the dependent variable was the effectiveness domain score and the independent variables were: age and gender (at enrollment), number of exacerbations, relevant spirometry parameters (Forced expiratory volume in the 1st second (FEV1) % of the predicted), level of dyspnea (MMRC score classes: 0-4), impact of COPD on a patient's life (CAT total score: 0-40) and treatment adherence (MMAS-4 score classes: 0-4) collected during observational period. Because dependent variable was collected at each study visit, repeated measures model was estimated taking into account all available values for dependent and independent variables.
  Mean is actually estimate of beta values. Visit 1 is at enrollment, visit 2 is at 6 months and visit 3 is at 12 months.
Time Frame: Up to 12 months
Population: FAS
Measure: Mean (Standard Error); unit: Beta coefficient estimate
Arm/Group | Total COPD Patients
Number analyzed (Participants) | 401
Beta coefficient estimate
  Visit 2 vs Visit 1 | 0.9639 (1.1450)
  Visit 3 vs Visit 1 | 1.8419 (1.2970)
  Age | -0.0566 (0.1015)
  Gender (Female vs Male) | 0.6152 (1.8658)
  Number of exacerbations in the year before Visit 1 | 0.1913 (1.0683)
  FEV1 predicted (%) at enrollment | 0.0924 (0.0387)
  MMAS-4 score class at Visit 1 (Score = 2 vs 4) | -1.7866 (2.1787)
  MMAS-4 score class at Visit 1 (Score = 3 vs 4) | -1.3991 (2.0051)
  CAT score at Visit 1 | -0.2645 (0.1137)
Statistical Analysis 1: Comparison: Total COPD Patients; Test type: Other; Intercept = 68.5027, Standard Deviation 8.0355 — Standard deviation is actually standard error

4. Secondary Outcome: The Relationship Between Treatment Satisfaction - Convenience Domain and Demographics, Clinical Parameters and Patient Reported Outcome (PROs) During a 12-month Observation Period.
Description: A regression model was estimated, where the dependent variable was the convenience domain score and the independent variables were: age and gender (at enrollment), number of exacerbations, relevant spirometry parameters (Forced expiratory volume in the 1st second (FEV1) % of the predicted), level of dyspnea (MMRC score classes: 0-4), impact of COPD on a patient's life (CAT total score: 0-40) and treatment adherence (MMAS-4 score classes: 0-4) collected during observational period. Because dependent variable was collected at each study visit, repeated measures model was estimated taking into account all available values for dependent and independent variables.
  Mean is actually estimate of beta values. Visit 1 is at enrollment, visit 2 is at 6 months and visit 3 is at 12 months.
Time Frame: Up to 12 months
Population: FAS
Measure: Mean (Standard Error); unit: Beta coefficient estimate
Arm/Group | Total COPD Patients
Number analyzed (Participants) | 401
Beta coefficient estimate
  Visit 2 vs Visit 1 | -0.1907 (1.0026)
  Visit 3 vs Visit 1 | 0.1130 (0.9902)
  Age | -0.2438 (0.0858)
  Gender (Female vs Male) | 0.1682 (1.5588)
  Number of exacerbations in the year before Visit 1 | -1.0434 (0.9070)
  FEV1 predicted (%) at enrollment | 0.0348 (0.0329)
  MMAS-4 score class at Visit 1 (Score = 2 vs 4) | -5.4461 (1.8328)
  MMAS-4 score class at Visit 1 (Score = 3 vs 4) | -4.2513 (1.6786)
  CAT score at Visit 1 | -0.0782 (0.0949)
Statistical Analysis 1: Comparison: Total COPD Patients; Test type: Other; Intercept = 95.4051, Standard Deviation 6.9951 — Standard deviation is actually standard error

5. Secondary Outcome: The Relationship Between Treatment Satisfaction - Global Satisfaction Domain and Demographics, Clinical Parameters and Patient Reported Outcome (PROs) During a 12-month Observation Period.
Description: A regression model was estimated, where the dependent variable was the global satisfaction domain score and the independent variables were: age and gender (at enrollment), number of exacerbations, relevant spirometry parameters (Forced expiratory volume in the 1st second (FEV1) % of the predicted), level of dyspnea (MMRC score classes: 0-4), impact of COPD on a patient's life (CAT total score: 0-40) and treatment adherence (MMAS-4 score classes: 0-4) collected during observational period. Because dependent variable was collected at each study visit, repeated measures model was estimated taking into account all available values for dependent and independent variables.
  Mean is actually estimate of beta values.Visit 1 is at enrollment, visit 2 is at 6 months and visit 3 is at 12 months.
Time Frame: Up to 12 months
Population: FAS
Measure: Mean (Standard Error); unit: Beta coefficient estimate
Arm/Group | Total COPD Patients
Number analyzed (Participants) | 401
Beta coefficient estimate
  Visit 2 vs Visit 1 | 2.2165 (1.0757)
  Visit 3 vs Visit 1 | 2.4258 (1.1032)
  Age | -0.1139 (0.1005)
  Gender (Female vs Male) | 1.6246 (1.8334)
  Number of exacerbations in the year before Visit 1 | -0.8055 (1.0599)
  FEV1 predicted (%) at enrollment | 0.0748 (0.0385)
  MMAS-4 score class at Visit 1 (Score = 2 vs 4) | -2.2278 (2.1607)
  MMAS-4 score class at Visit 1 (Score = 3 vs 4) | -5.4749 (1.9726)
  CAT score at Visit 1 | -0.2445 (0.1117)
Statistical Analysis 1: Comparison: Total COPD Patients; Test type: Other; Intercept = 74.8895, Standard Deviation 8.0048 — Standard deviation is actually standard error

6. Secondary Outcome: The Health Care Resources Utilization According to the Italian National Health Service (INHS) During a 12-month Observation Period
Description: Health care resources consumption related to COPD, COPD exacerbations and COPD-drug-related adverse events was computed during observational period in terms of number of (inward and day-hospital) hospitalizations, number of emergency room accesses, number of General Practitioner (GP) visits, specialist visits and laboratory tests or examinations.
  Hospitalization (Number Analyzed) - Number of hospitalizations not in ICU during observation period per patient, Emergency room accesses (Number Analyzed) - Number of Emergency room accesses during observation period per patient, Specialist Outpatient Visits (Number Analyzed) - Number of specialist outpatient visits per patient during observation period, GP Visits (Number Analyzed) - Number of general practitioner visits per patient during observation period, Laboratory Tests (Number Analyzed) - Number of tests per patient during observation period.
Time Frame: Up to 12 months
Population: FAS
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Total COPD Patients
Number analyzed (Participants) | 401
Number of events
  Hospitalization | 0.1 (0.4)
  Emergency room accesses | 0.1 (0.2)
  Specialist Outpatient Visits | 0.2 (0.7)
  GP Visits | 0.4 (0.9)
  Laboratory Tests | 0.7 (3.1)

7. Secondary Outcome: Correlation Between Patients' Satisfaction and Resource Utilization
Description: Correlation indexes were calculated between treatment satisfaction domain scores of TSQM-9 and healthcare resource consumption at 12-month follow-up visit.
  Hospitalization - Number of hospitalizations not in ICU during observation period per patient, Specialist Outpatient - Number of specialist outpatient visits per patient during observation period, E = Effectiveness at 12 months and C = Convenience at 12 months
Time Frame: 12-month follow-up visit
Population: FAS
Measure: Number; unit: Spearman's correlation coefficients
Arm/Group | Total COPD Patients
Number analyzed (Participants) | 401
Spearman's correlation coefficients
  Specialist Outpatient_E: number analyzed (Participants) | 304
  Specialist Outpatient_E | -0.14945
  Hospitalization_C: number analyzed (Participants) | 304
  Hospitalization_C | -0.13233

ADVERSE EVENTS:
Time Frame: From signing the informed consent till the end of the study (Visit3 after 12 months +/- 1 months).
Arm/Group | Total COPD Patients
All-Cause Mortality (participants affected / at risk) | 9/401
Serious Adverse Events (participants affected / at risk) | 12/401
Other Adverse Events (participants affected / at risk) | 0/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total COPD Patients (N=401)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Death (General disorders) | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sudden cardiac death (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Neither study was designed to prove the existence clinical factors of any causal relationship nor foreseen a selection method for balanced groups. Neither treatment satisfaction was assessed nor validated to identify patients' satisfaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-07-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02689492/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT02689492/SAP_001.pdf